CLINICAL TRIAL: NCT05170308
Title: Fractional CO2 Laser for the Treatment of Lichen Planus Pigmentosus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient patient population to enroll
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Heather Woodworth Goff, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2021-0551
Record Dates: First submitted 2021-12-08; First posted 2021-12-27 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Lichen Planus Pigmentosus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment (CO2 fractional laser) arm (Other): CO2 fractional laser will be used to treat dyspigmentation in lichen planus pigmentosus in one half along sagittal midline section in each subject.
  Interventions: Device: CO2 fractional laser
- No treatment (Control) arm (No Intervention): One half along sagittal midline section in each subject will not receive the CO2 fractional laser treatment.

INTERVENTIONS:
Device: CO2 fractional laser — The study subjects' body will be divided into two equal halves along sagittal midline section with one side receiving treatment with fractional CO2 laser (experimental) to treat dyspigmentation in lichen planus pigmentosus
  Other Names: SmartXide DEKA DOT
  Arms: Treatment (CO2 fractional laser) arm

SUMMARY:
This study will assess the safety and efficacy of fractional carbon dioxide (CO2) laser treatment for Lichen Planus Pigmentosus (LPP). LPP is a chronic pigmentary disorder typically involving the forehead, lateral cheeks, and occasionally other sun-exposed areas such as the forearms. Clinically, LPP appears as a reticulated brown to black macules and patches. Previously studied effective treatments of LPP include topical tacrolimus and corticosteroids. LPP is often recalcitrant to therapy, with chronic maintenance treatment needed to prevent repigmentation. There are few reports of laser modalities being used to treat LPP, with Nd:YAG being the only published laser modality to be attempted. Although topical therapies are relatively safe, there is a lack of satisfactory treatment options for this patient population. Fractional CO2 laser has been widely used for photoaging due to its effectiveness and high safety profile. Clinically evident improvement can be appreciated even after only one session of treatment.

Ablative fractional laser resurfacing is both safe and effective for the treatment of the vascular, pigmentary and textural components of skin disorders. No data exist regarding the use of fractional CO2 laser for management of LPP. This study hopes to fulfill this purpose.

The study subjects' body will be divided into two equal halves along sagittal midline section with one side receiving treatment with fractional CO2 laser (experimental) and the other left untreated (control)

DETAILED DESCRIPTION:
Patients with a clinical diagnosis of LPP defined by a skin biopsy will be recruited. Ten patients will be consented. Before the initial visit, all patients will complete a one-month preoperative daily use of SPF 50+ sunscreen. The sun protection is to reduce further sun damage and protect skin from increased photosensitivity that may occur after laser resurfacing. At the initial visit, high resolution photographs of the affected area will be taken. All patients in each group will fill out a form with demographic information. Patients will be instructed to come to their appointment with clean skin and without any lotions or moisturizers on the area. Laser-specific eyewear will be provided to practitioners, patients, and all other people in the treatment room. A blue skin marking pen will be used to draw a line separating the body into two equal halves. Compounded benzocaine, lidocaine, and tetracaine (BLT) cream in a 20:8:4% concentration will be applied to the treatment area for 40 minutes prior to the procedure. Before the treatment, topical anesthesia will be thoroughly washed off with chlorhexidine gluconate and distilled water. One pass with a 1-mm spot density and a 60micron depth will be performed followed by a 1mm spot density and a 200-micron depth will be used. The left half of the testing area will be left intact and used as the control for easy comparison. Forced cold air (Zimmer cooler) will also be used in conjunction with the laser device for better patient comfort.

Cold compresses with refrigerated distilled water can be used to reduce swelling and to soothe the skin with frequent reapplication of white petrolatum to keep the skin coated for days 1-5 post-procedure with strict sun avoidance for the first week post-procedure. Daily use of broad-spectrum sunscreen with SPF50+ will be required after the first week.

Given the current pandemic, limited in-person follow-ups will be scheduled (once at baseline before treatment, then at 12 and 24-weeks post-treatment. Participants will communicate immediate post-treatment issues or concerns along with selfies through MyChart on day 2, 3, 7, 10, 14 to track progress and to identify any post procedural complications in a timely fashion.

There will also be no costs to the patients for the laser procedures as funding will be supplied by the UT Southwestern Dermatology department via an educational grant. Patients desiring treatment of the control side after the study end-point (24 weeks) will be provided at no cost for the participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, English and non-English speakers, and subjects more than 18 years old
* Histologic diagnosis of LPP affecting the bilateral body
* Willing to refrain from using other topical medications other than the topical medications provided to patients.
* Agree to not undergo any other procedures on affected area during the study
* Agree to refrain from tanning for 6 months post-procedure
* Willing and able to read, understand, and sign the consent form
* Willing and able to adhere to the treatment and follow-up schedule as well as post-treatment care

Exclusion Criteria:

* Patients under 18 years old
* Active skin infection, dermatitis, or a rash on the treatment area
* Pregnant or lactating patients
* Patients on immunosuppressive medications
* Any laser procedures or chemical peel procedures on the affected area within the past 6 months
* Patients with multiple comorbidities such as diabetes mellitus, cardiovascular diseases, neurologic disorders, internal malignancies
* Personal history or family history of forming keloids or hypertrophic scars, or abnormal wound healing
* Patients with known bleeding disorders or taking more than one anticoagulation medications
* Undergoing any surgery in the treatment area within the past 12 months
* History of radiation to the head, neck, and chest area
* Systemic use of isotretinoin within 6 months
* Any use of gold therapy
* Current smoker or history of smoking within 12 months of study
* ny physical or mental condition in which the investigators deem unsafe for the subject to participate in the study.
* History of recurrent herpes simplex on the affected area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in dyspigmentation at 12 weeks post treatment | 12 weeks post treatment
  Improvement in dyspigmentation at 12 weeks post treatment is assessed by the Physician's Global Aesthetic Improvement Scale which is a 11-point scale. Each dermatologist from an independent panel (blinded to treatment parameters and the treatment laterality at each photograph time point) will be asked to identify the baseline and post-treatment images from randomized, paired images for all subjects. Reviewers will rate improvement in LPP in 10% increments on an 11-point scale (0% no improvement to 100% or complete clearance).
Improvement in dyspigmentation at 24 weeks post treatment | 24 weeks post treatment
  Improvement in dyspigmentation at 24 weeks post treatment is assessed by the Physician's Global Aesthetic Improvement Scale which is a 11-point scale. Each dermatologist from an independent panel (blinded to treatment parameters and the treatment laterality at each photograph time point) will be asked to identify the baseline and post-treatment images from randomized, paired images for all subjects. Reviewers will rate improvement in LPP in 10% increments on an 11-point scale (0% no improvement to 100% or complete clearance).

SECONDARY OUTCOMES:
Overall Subject Satisfaction assessed at 12 weeks post treatment | 12 weeks post treatment
  Overall Subject Satisfaction with improvement of LPP is assessed at 12 weeks post treatment using an 5-point satisfaction and aesthetic scale. Possible scores range from 0-5, where higher scores indicate better outcome.
Overall Subject Satisfaction assessed at 24 weeks post treatment | 24 weeks post treatment
  Overall Subject Satisfaction with improvement of LPP is assessed at 24 weeks post treatment using an 5-point satisfaction and aesthetic scale. Possible scores range from 0-5, where higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Goff, MD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No